CLINICAL TRIAL: NCT01444807
Title: A Randomized, Open Label, Multicenter Phase 2 Study, to Evaluate the Efficacy of Sorafenib in Patients With Advanced Renal Cell Carcinoma (RCC) After a Radical Resection of the Metastases
Brief Title: Evaluate the Efficacy of Sorafenib in Renal Cell Carcinoma Patients After a Radical Resection of the Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: GP1
Record Dates: First submitted 2011-09-08; First posted 2011-10-03 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: sorafenib; metastatic renal cell carcinoma; metastasectomy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib (Experimental): Active Arm
  Interventions: Drug: sorafenib
- Best Supportive Care (No Intervention): Comparator

INTERVENTIONS:
Drug: sorafenib — sorafenib 400 mg bid
  Other Names: Nexavar (Bayer Health Care - Leverkusen - Germany)
  Arms: Sorafenib

SUMMARY:
Evaluate the efficacy and tolerability of sorafenib in RCC patients underwent to metastasectomy

DETAILED DESCRIPTION:
Advanced RCC presents poor prognosis, because its pathogenesis is not clearly understood. However, up-regulation of the Ras pathway is thought to play a role.

VEGF expression could represent independent prognostic factors for survival possibly linking expression of this protein with clinical outcome.

Sorafenib is a potent inhibitor of both Raf-kinase and VEGF R2 signalling The anti-tumoral activity of Sorafenib was clearly demonstrated in phase III trial regarding advanced pretreated RCC.

Surgical removal of metastatic disease could potentially increase the disease control rate.

Particularly in patients with a disease free interval post nephrectomy of at least 1 year, with one small metastatic lesion, metastasectomy could represents an important therapeutic approach.

After a radical resection of the metastatic disease is unclear if an anti-tumoral systemic therapy may increase patient survival.

In summary, both the preclinical and clinical data support further evaluation of Sorafenib in RCC patients.

ELIGIBILITY:
INCLUSION CRITERIA

* Age ≥ 18 years
* Patients with cytological or histological diagnosis of Renal Cell Carcinoma (RCC)
* Absence of residual lesions following surgical removal of metastatic disease. Assessment must be performed by CT-scan or MRI
* Histologically proven disease free margins of resected surgical specimen
* No more than three months from radical resection on metastases.
* ECOG Performance Status of 0 or 2
* Life expectancy of at least 12 weeks.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:
* Hemoglobin > 9.0 g/dl
* Absolute neutrophil count (ANC) >1,500/mm3
* Platelet count 100,000/ml
* Total bilirubin < 1.5 times the upper limit of normal
* ALT and AST < 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer)
* Alkaline phosphatase 4 x ULN
* PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.] For patients on warfarin, close monitoring of at least weekly evaluations will be performed, until INR is stable based on a measurement at pre-dose, as defined by the local standard of care.
* Serum creatinine < 1.5 x upper limit of normal
* Amylase and lipase <1.5 X upper limit of normal
* Signed informed consent must be obtained prior to any study specific procedures

EXCLUSION CRITERIA:

* Prior systemic treatment for metastatic RCC. It is allowed an adjuvant or neoadjuvant therapy before or after nephrectomy if stopped at least 6 months before the resection of metastatic lesion/s.
* History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 mo prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension (>= 160 mmHg systolic and/or 90 mmHg diastolic).
* History of HIV infection or chronic hepatitis B or C
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry. Also the patient must not be undergoing acute steroid therapy or taper (chronic steroid therapy is acceptable provided that the dose is stable for one month prior to and following screening radiographic studies)
* Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
* History of organ allograft
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* History of other disease, metabolic dysfunction, physical examination finding or clinical laboratory finding giving reasonable suspicion of a disease condition that contraindicates use of an investigational drug or patient at high risk from treatment complications
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1) or any cancer curatively treated > 3 years prior to study entry.
* Anticancer chemotherapy or immunotherapy during the study or within 4 weeks of study entry.
* Radiotherapy during study or within 3 weeks of start of study drug.
* Major surgery within 4 weeks of start of study
* Autologous bone marrow transplant or stem cell rescue within 4 months of study
* Use of biologic response modifiers, such as G-CSF, within 3 week of study entry. (G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator, however they may not be substituted for a required dose reduction.) (Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study)
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry
* Prior exposure to the study drug.
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and two weeks after the completion of trial.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
* Patients unable to swallow oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-03 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival | December 2011 - December 2014 (3 years)
  Efficacy of Sorafenib compared with BSC, in RCC patients that have undergone radical resection of recurrent metastatic disease, after prior nephrectomy. The primary efficacy endpoint is Recurrence Free Survival (RFS),

SECONDARY OUTCOMES:
Overall Survival | December 2011 - December 2014 (3 years)
Safety Profile | December 2011 - December 2014 (3 years)
  Physical examination, vital signs, Red blood count: haemoglobin, hematocrit, platelet count, white blood cell count. WBC should include differential neutrophil, lymphocyte, monocyte, basophil and eosinophil counts. Electrolyte panel: sodium, potassium, chloride and corrected calcium.Chemistry panel: AST, ALT, bilirubin, alkaline phosphatase, uric acid, total protein, albumin, calcium, lipase, amylase, phosphate, LDH, glucose, creatinine,BUN, and bicarbonate. Coagulation panel: PT, PT-INR, PTT. Urinalysis, Adverse event
Vascular endothelial growth factors (VEGF) levels in BSC and Sorafenib arm. | December 2011 - December 2014 (3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Procopio, MD, Study Chair — Istituto Tumori Milano
Locations (14):
- Italy (14):
  - Istituto Tumori Milano, Milan, Mi
  - Cinzia Ortega, Alba
  - Alessandra Bearz, Aviano
  - Alfredo Berruti, Brescia
  - Saverio Cinieri, Brindisi
  - Francesco Atzori, Cagliari
  - Rodolfo Passalaqua, Cremona
  - Francesco Di Costanzo, Florence
  - Vincenzo Emanuele Chiuri, Lecce
  - Alessandra Mosca, Novara
  - Vittorio Gebbia, Palermo
  - Enrico Cortesi, Roma
  - Francesco Cognetti, Roma
  - Franco Morelli, San Giovanni Rotondo

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ljungberg B. The role of metastasectomy in renal cell carcinoma in the era of targeted therapy. Curr Urol Rep. 2013 Feb;14(1):19-25. doi: 10.1007/s11934-012-0293-6. PMID 23212738